CLINICAL TRIAL: NCT02257541
Title: A Phase Ib/II Study of BGJ398 in Combination With Imatinib Mesylate in Patients With Untreated Advanced Gastrointestinal Stromal Tumor (GIST)
Brief Title: BGJ398 in Combination With Imatinib Mesylate in Patients With Untreated Advanced Gastrointestinal Stromal Tumor (GIST)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Dana-Farber Cancer Institute (Other); M.D. Anderson Cancer Center (Other); University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-140
Record Dates: First submitted 2014-10-02; First posted 2014-10-06 (Estimated); Results first posted 2020-03-30 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2019-03

CONDITIONS: Advanced Gastrointestinal Stromal Tumor (GIST)
Keywords: BGJ398; Imatinib Mesylate; 14-140
MeSH Terms: interventions — infigratinib; Imatinib Mesylate

ARMS (1):
- BGJ398 With Imatinib Mesylate (Experimental): BGJ398 With Imatinib Mesylate In the phase Ib portion of the study, patients will receive imatinib at 400 mg once daily and BGJ398 at the standard 3+3 escalation doses for 21 days on, 7 days off (treatment schedule A).Using treatment schedule A, if dose level 1 to -2 is identified as the MTD and concern exists regarding therapeutic activity of BGJ398 at this dose level, expansions with higher dose levels (1 to 3) may be considered at the MSKCC PI's discretion, with modification of the treatment schedule. In this setting BGJ398 will be administered daily for one week followed by 3 weeks off and imatinib will be taken daily throughout the 4 week cycle period (treatment schedule B). In the phase II portion of the study, patients will receive imatinib at 400 mg once daily (standard of care first line imatinib dose) and BGJ398 at the RP2D and treatment schedule identified in the phase Ib portion of the study. One cycle is 28 days.
  Interventions: Drug: BGJ398; Drug: Imatinib Mesylate

INTERVENTIONS:
Drug: BGJ398
Drug: Imatinib Mesylate

SUMMARY:
The goal of a phase Ib clinical trial is to find the doses of drugs that are safe. Although BGJ398 has been given to patients safely on its own, it has never been given together with imatinib mesylate. In this study, we will test the safety of taking BGJ398 with imatinib mesylate. The investigators will learn this by closely checking for side effects that the patient may experience. Side effects can be seen in laboratory studies, on physical examination, or by asking the patient.Once a dose has been determined to be safe, a larger Phase II study will be done in patients with advanced GIST who have never received any prior treatments.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pathologically confirmed GIST.
* In the Phase Ib portion, must have locally advanced or metastatic GIST and have progressed on imatinib.
* In the Phase II portion, patients must be newly diagnosed or imatinib treatment naïve in the advanced/metastatic setting. Prior adjuvant imatinib therapy is allowed as long as disease recurrence was documented ≥90 days after last dose of imatinib and imatinib has not yet been restarted.
* Patients must be at least 18 years of age.
* Disease must be measurable by RECIST 1.1.
* ECOG Performance Status 0 or 1. Adequate renal, hepatic, and hematologic function as the following: Serum Creatinine ≤ 1.5 mg/dL, Total Serum Bilirubin ≤ 1.5 x upper limit of normal (ULN) unless due to Gilbert's Disease, Serum AST (SGOT) and/or ALT (SGPT) ≤ 2.5 x ULN (or ≤ 5.0 x ULN if considered due to tumor), ANC ≥ 1500/mm3, Platelets ≥ 100,000/mm3, and hemoglobin ≥ 10g/dL.
* Patients of childbearing potential must have a negative blood pregnancy test within 14 days of treatment. Patients must agree to use a reliable barrier method of birth control during and for 3 months following the last dose of study drug.
* Patient must have adequate cardiac function (left ventricular ejection fraction (LVEF) ≥50% as determined by a multigated acquisition (MUGA) scan or echocardiogram; and QTc interval ≤480 ms by Fridericia's formula (QTcF).
* Patient must be able to take oral medications.
* Patients must sign an informed consent document.

Exclusion Criteria:

* For phase I, prior intolerance to imatinib at a dose of 400 mg daily.
* For phase II, any receipt of cytotoxic, biologic, or immune therapy aimed to treat GIST except for adjuvant imatinib systemic therapy that concluded at least 90 days prior to registration. For Phase I, patients are eligible regardless of prior therapy.
* Chronic liver disease (e.g., cirrhosis)
* Known positive serology for HIV, active Hepatitis B, and/or active Hepatitis C infection.
* Patients have a history or current evidence of Central Serous Retinopathy (CSR) or retinal vein occlusion (RVO) or major predisposing factors to CSR or RVO (e.g. uncontrolled glaucoma or ocular hypertension) in the opinion of the study ophthalmologist.
* History of retinal degenerative disease
* Active corneal disorder or keratopathy (e.g. corneal abrasion, bullous keratopathy)
* Severe and/or uncontrolled medical disease, including:

  * Uncontrolled diabetes mellitus (A1c >8)
  * Chronic Kidney Disease Stage III or higher (Creatinine Clearance <60mL/min/m2 by Modified Diet in Renal Disease (MDRD) calculation)
  * Active, uncontrolled infection Known active brain metastasis unless they have been treated and shown documented radiographic stability for 28 days.
* Known other active malignancy (other than malignancies which the investigator determines are unlikely to interfere with treatment and safety analysis).
* Patients have clinically significant cardiovascular disease, including any of the following

  * Any history of acute coronary syndrome including myocardial infarction, stable or unstable angina, CABG, coronary angioplasty or stenting or known obstructive coronary artery disease.
  * Symptomatic chronic heart failure (New York Heart Association Criteria, Class II-IV)
  * Evidence of clinically significant cardiac arrhythmias and/or conduction abnormalities < 6 months prior to screening except atrial fibrillation (AF) and paroxysmal supraventricular tachycardia (PSVT)
* Any history of thrombotic cerebrovascular accident or other arterial thrombosis
* Uncontrolled arterial hypertension (systolic blood pressure >155 mmHg or diastolic >95 mmHg) despite appropriate medical therapy.
* History and/or current evidence of uncontrolled endocrine alterations of calcium/phosphate homeostasis, e.g., parathyroid disorders, history of parathyroidectomy, tumor lysis, tumoral calcinosis, etc.
* Impairment of gastrointestinal function or gastrointestinal disease (e.g., uncontrolled ulcerative disease; uncontrolled nausea, vomiting, diarrhea; chronic malabsorption syndrome).
* Patients with major surgery within 3 weeks prior to study entry or who have not recovered from side effects of such procedure.
* Women who are pregnant or lactating.
* Sexually active males, unless they use a condom during intercourse while taking the drug and for 15 days after stopping treatment. They should not father a child in this period. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid.
* Patients with any significant history of non-adherence to medical regimens or with inability to grant reliable informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-10-02 (Actual); Primary Completion 2019-03-25 (Actual); Study Completion 2019-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Tap, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memoral Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering at Mercy Medical Center, Rockville Centre, New York
  - Md Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Kelly CM, Shoushtari AN, Qin LX, D'Angelo SP, Dickson MA, Gounder MM, Keohan ML, Mcfadyen C, Sjoberg A, Singer S, DeMatteo RP, Hwang S, Heinemann MH, Francis JH, Antonescu CR, Chi P, Tap WD. A phase Ib study of BGJ398, a pan-FGFR kinase inhibitor in combination with imatinib in patients with advanced gastrointestinal stromal tumor. Invest New Drugs. 2019 Apr;37(2):282-290. doi: 10.1007/s10637-018-0648-z. Epub 2018 Aug 13. PMID 30101387
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1b, Dose Level -1: Phase 1b, Dose Level -1: BGJ398 50 mg
- Phase 1b, Dose Level 1: Phase 1b, Dose Level 1: BGJ398 75 mg
- Phase 1b, Dose Level 2: Phase 1b, Dose Level 2: BGJ398 100 mg
- Phase 1b, Dose Level -2: Phase 1b, Dose Level -2: BGJ398 25 mg
- Phase II: Phase II: BGJ398 75mg
Period: Overall Study
Arm/Group | Phase 1b, Dose Level -1 | Phase 1b, Dose Level 1 | Phase 1b, Dose Level 2 | Phase 1b, Dose Level -2 | Phase II
Started | 3 | 8 | 1 | 3 | 1
Completed | 3 | 8 | 1 | 3 | 1
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1b, Dose Level -1 | Phase 1b, Dose Level 1 | Phase 1b, Dose Level 2 | Phase 1b, Dose Level -2 | Phase II | Total
Number analyzed (Participants) | 3 | 8 | 1 | 3 | 1 | 16
Age, Continuous [Median (Full Range); unit: years] | 54 [48 to 65] | 58.88 [47 to 77] | 44 [44 to 44] | 53 [49 to 64] | 53 [53 to 53] | 54 [44 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 0 | 0 | 1 | 3
  Male | 3 | 6 | 1 | 3 | 0 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 3 | 6 | 0 | 3 | 0 | 12
  Unknown or Not Reported | 0 | 1 | 1 | 0 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 0 | 0 | 2
  White | 2 | 4 | 1 | 3 | 0 | 10
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 8 | 1 | 3 | 1 | 16

OUTCOME MEASURES:

1. Primary Outcome: Phase Ib Study: Number of Participants With Dose-Limiting Toxicities
Description: The phase Ib will be pursued in standard 3+3 format, based on toxicities encountered during the first cycle of therapy.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b, Dose Level -1 | Phase 1b, Dose Level 1 | Phase 1b, Dose Level 2 | Phase 1b, Dose Level -2
Number analyzed (Participants) | 3 | 8 | 1 | 3
Participants | 3 | 8 | 1 | 3

2. Primary Outcome: Phase Ib Portion: Response Rate (RR)
Description: (CR+PR, RECIST 1.1) and by CHOI criteria
  PHASE 1b PARTICIPANTS ONLY
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: 32 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b, Dose Level -1 | Phase 1b, Dose Level 1 | Phase 1b, Dose Level 2 | Phase 1b, Dose Level -2
Number analyzed (Participants) | 3 | 8 | 1 | 3
Participants
  Partial Response/PR | 1 | 0 | 0 | 0
  Stable Disease/SD | 2 | 3 | 0 | 0
  Progressive Disease/PD | 0 | 3 | 1 | 3
  Not reported due to withdrawn from study | 0 | 2 | 0 | 0

3. Secondary Outcome: Phase Ib Study: Response Rate (RR)
Description: defined by RECIST 1.1 criteria and by CHOI criteria,and by EORTC criteria
  PHASE 1b PARTICIPANTS ONLY
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: 32 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b, Dose Level -1 | Phase 1b, Dose Level 1 | Phase 1b, Dose Level 2 | Phase 1b, Dose Level -2
Number analyzed (Participants) | 3 | 8 | 1 | 3
Participants
  Progressive Disease/PD | 1 | 2 | 0 | 3
  Stable Disease/SD | 2 | 4 | 1 | 0
  Not reported due to withdrawn from study | 0 | 2 | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Phase 1b, Dose Level 2:: Phase 1b, Dose Level 2: BGJ398 100 mg
Arm/Group | Phase 1b, Dose Level -1 | Phase 1b, Dose Level 1 | Phase 1b, Dose Level 2: | Phase 1b, Dose Level -2 | Phase II
All-Cause Mortality (participants affected / at risk) | 2/3 | 3/8 | 0/1 | 0/3 | 0/1
Serious Adverse Events (participants affected / at risk) | 2/3 | 7/8 | 1/1 | 3/3 | 0/1
Other Adverse Events (participants affected / at risk) | 3/3 | 8/8 | 1/1 | 3/3 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b, Dose Level -1 (N=3) | Phase 1b, Dose Level 1 (N=8) | Phase 1b, Dose Level 2: (N=1) | Phase 1b, Dose Level -2 (N=3) | Phase II (N=1)
CPK increased (Investigations) | 1 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Intra-Abdominal Bleeding (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Ejection Fraction decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Lipase Increased (Investigations) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b, Dose Level -1 (N=3) | Phase 1b, Dose Level 1 (N=8) | Phase 1b, Dose Level 2: (N=1) | Phase 1b, Dose Level -2 (N=3) | Phase II (N=1)
Abdominal pain (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 1
Anemia (Blood and lymphatic system disorders) | 3 | 3 | 1 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
AST Elevated (Investigations) | 1 | 0 | 0 | 2 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0
Chest Pain - Cardiac (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 3 | 1 | 0 | 0
CPK Increased (Investigations) | 3 | 4 | 0 | 1 | 1
Creatinine Increased (Investigations) | 1 | 1 | 0 | 0 | 0
Decreased TSH (Investigations) | 1 | 0 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 3 | 0 | 0 | 0
Dry Mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Edema Limbs (General disorders) | 1 | 1 | 0 | 1 | 0
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 | 0 | 1 | 1 | 1
Fatigue (General disorders) | 2 | 5 | 0 | 0 | 0
Flashing Lights (Eye disorders) | 1 | 0 | 0 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hyperphosphatemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 2 | 1 | 1 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 0 | 0
Lipase Increased (Investigations) | 2 | 3 | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0
Pain (General disorders) | 1 | 0 | 1 | 0 | 0
Sleep Apnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1 | 0 | 0
Alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Anorexia (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Bloating (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blurred Vision (Eye disorders) | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Dry Eye (Eye disorders) | 0 | 2 | 0 | 0 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 2 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Memory Impairment (Nervous system disorders) | 0 | 2 | 0 | 0 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 0
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Serum amylase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Weight gain (Investigations) | 0 | 1 | 0 | 0 | 0
Weight loss (Investigations) | 0 | 1 | 0 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 1 | 1 | 0
Fever (General disorders) | 0 | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Periorbital edema (Eye disorders) | 0 | 0 | 0 | 1 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 1
Watering eyes (Eye disorders) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-24): https://cdn.clinicaltrials.gov/large-docs/41/NCT02257541/Prot_SAP_000.pdf